CLINICAL TRIAL: NCT04259762
Title: Enhancing Cancer Prevention and Control Pathways-Native Health Initiative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: University of New Mexico (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 18-264; P20GM103451 (NIH)
Record Dates: First submitted 2020-01-30; First posted 2020-02-06 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-03

CONDITIONS: Cancer, Breast; Cancer, Colon; Cancer, Cervix
Keywords: breast neoplasm; colorectal neoplasm; cervical neoplasm; screening; behavioral interventions; American Indians
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Enrollment numbers for Aims 3 and 4 are 96 and 281, respectively. The enrollment number n=131 is for Aim 8, INT, Pilot Test only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aim 8 (INT, Pilot Test): Breast, Colorectal, and Cervical Cancer Screening (Experimental): The study staff will administer to eligible participants the pre-INT and post-INT surveys. The post-INT surveys will be administered approximately 8 months after delivering the INTs. The participants will receive the INT(s) immediately after completing the pre-INT surveys.
  Interventions: Other: Aim 8 (INT, Pilot Test): Breast, Colorectal, and Cervical Cancer Screening Cognitive-Behavioral Interventions

INTERVENTIONS:
Other: Aim 8 (INT, Pilot Test): Breast, Colorectal, and Cervical Cancer Screening Cognitive-Behavioral Interventions — Adult men and women will receive age- and gender-specific INTs. Women age 45-75 years will receive the interventions for breast, colorectal, and cervical cancers screening. Men age 45-75 years will receive the intervention for colorectal cancer screening. Women age 21-49 years will receive the intervention for cervical cancer screening. The cognitive-behavioral INTs on age-gender specific cancers will range from 1-2 hours. The study team will utilize a digital flipchart that will cover each cancer's specific risk/protective factors, incidence, mortality, screening methods, and resources. The study team member delivering the INTs will function as a facilitator linking information with practical skills.

SUMMARY:
There are continued disparities in cancer incidence, mortality, and survival between American Indians (AIs) and Whites on cancers responsive to early screening (i.e., breast, colorectal, and cervical) in the US. In New Mexico (NM), AIs compared with other racial/ethnic populations are significantly less likely to adhere to recommended screening guidelines. The purpose of this trial is to develop and pilot test multilevel/multicomponent intervention strategies to enhance screening for breast, colorectal, and cervical cancers.

DETAILED DESCRIPTION:
There are continued disparities in cancer incidence, mortality, and survival between American Indians (AIs) and Whites on cancers responsive to early screening (i.e., breast, colorectal, and cervical) in the US. Between 1990-2009, based on data from Contract Health Service Delivery Area Counties across the US, the mortality-to-incidence ratios for these cancers were significantly higher for American Indian/Alaska Natives compared to Whites (breast: 1.22, colorectal: 1.16, cervix: 1.36), indicating poorer survival. New Mexico (NM) AIs also experience substantial cancer disparities. Between 2010-2014, AIs compared to Whites had higher incidence (per 100,000) for cervical (7.9 vs. 6.9) and colorectal (male: 46.5 vs. 35.2; female: 29.2 vs. 28.2) cancers, and higher mortality for cervical (3.7 vs. 1.3) and colorectal (males only; 18.9 vs. 15.6) cancers. AIs were more likely to receive a late-stage (i.e., regional or distant) cancer diagnosis for all 3 screen detectable cancers. AIs have some of the lowest cancer screening rates compared with other racial/ethnic groups. In NM, AIs listed in the Indian Health Service (IHS) Albuquerque Area have substantially lower screening rates than the state's White population do. AIs had screening rates of: breast (58.5%, women ages 52-64), colorectal (41.9%, ages 50-75), and cervical (63.9%, women ages 24-64) cancers; whereas, screening rates for Whites were: breast (70.0%, ages 50-74), colorectal (69.2%, ages 50-75), and cervical (77.8%, women 21-65)

The overall objective is to develop and pilot test culturally and linguistically appropriate interventions to enhance age- and risk-appropriate breast, colorectal, and cervical cancer screening in concordance with the U.S. Preventive Services Task Force recommended guidelines

Aim 3 (Focus Groups, Descriptive): Qualitative documentation of perspectives on cancer control needs in the Zuni Pueblo

Protocol: Aim 3 (Focus Groups, Descriptive): Qualitative documentation of perspectives on cancer control needs in the Zuni Pueblo

1. Research Design: Focus groups that gather qualitative (descriptive) perspectives and insights from a small group of participants
2. Research Setting: Zuni Pueblo
3. Participant identification and sampling: Non-probability sampling
4. Procedures: The investigators will contact interested participants for focus group sessions
5. Primary Outcome: Knowledge about, barriers and support for, and communication about breast, cervix, and colorectal cancers
6. Data Analysis: Thematic analyses of transcripts of the focus group discussions
7. Sample Size Considerations: The investigators will enroll about 8-10 participants per focus group

Aim 4 (Community Survey, Descriptive): Documentation of perspectives on cancer control needs in the Zuni Pueblo

Protocol: Aim 4 (Community Survey, Descriptive): Documentation of perspectives on cancer control needs in the Zuni Pueblo

1. Research Design: Cross-sectional
2. Research Setting: Zuni Pueblo
3. Participant identification and sampling: The sampling strategy for the Community Survey includes random sampling of streets, strategic convenience sampling, and snowball sampling.
4. Procedures: The investigators will implement the Community Survey among interested and eligible participants. Participants will complete surveys documenting cancer control needs for breast, cervix, or colorectal cancers. Women aged 50-75 will be surveyed on breast, cervix, and colorectal cancers; women aged 21-49 will be surveyed on cervix cancer, and men aged 50-75 will be surveyed on colorectal cancer
5. Primary Outcome: Self-reported screening behaviors for breast, colorectal, and cervix cancers
6. Data Analysis: Descriptive analysis of survey data
7. Sample Size Considerations: The investigators will enroll about 300 participants

Aim 8 (INT, Pilot Test). Pilot test multilevel/multicomponent interventions on screening outcomes

Protocol. Aim 8 (INT, Pilot Test): Pilot Test Effectiveness of the Multilevel/Multicomponent Intervention [INT]

1. Research Design: One-group, pre-INT/post-INT
2. Research Setting: Zuni Pueblo
3. Randomization: Non-randomized, convenience sampling
4. Participant Identification and Sampling: The investigators will identify and contact participants who had previously expressed interest in participating in the pilot testing of any of the 3 cancer-specific INTs
5. Interventions: Educational and behavioral INTs on cancers of the breast, colorectal, and cervix
6. Procedures: The investigators will contact interested participants and redetermine eligibility. Eligible participants will complete baseline (pre-INT) and post-INT surveys about 6-8 months after receiving the INT(s). The surveys will be administered in-person or over the phone and will last approximately 20-30 minutes
7. Implementation of the INTs: The investigators could operationalize recommended strategies that may plausibly include strategies to: To increase community access, the investigators could: (a) Identify a point-person at the health center who will triage participants to and schedule them for appropriate screening(s). (b) Remind participants to complete their screening exam(s), offer assistance in scheduling a screening appointment and a ride to the health center. These strategies would reduce administrative barriers, navigate participants, and assist with transportation and in scheduling an appointment. To increase community demand, the investigators could consider: (a) Educational materials. (b) 1-on-1 education. (c) Cognitive-behavioral group education and incentives. To increase provider delivery, the investigators could: (a) Reduce health center-specific systemic barriers by identifying a point-person to promote and facilitate screening services
8. Baseline and Post-intervention Surveys: The investigators will collect data on demographics, self-reported receipt of a cancer-specific screening exam, self-reported scheduling of an appointment to obtain a cancer-specific screening exam, or self-reported attempt to make an appointment for a cancer-specific screening exam
9. Primary Outcome: Self-reported receipt of a screening exam, or scheduling an appointment for a screening exam, or self-reported attempt to make an appointment for a screening exam. Cancer-specific screening exams include FOBT/FIT/Colonoscopy for colorectal cancer, Pap smear for cervical cancer, or mammogram for breast cancer
10. Data Analysis: The investigators will compute the count of participants who self-reported receipt of a screening exam, scheduling an appointment for a screening exam, or attempt to make an appointment for a screening exam. These analyses will be presented by age/sex strata. Men age 45-75 for colorectal cancer screening; women 45-75 for breast, cervical, and colorectal cancer screening; and women 21-49 for cervical cancer screening
11. Sample Size Considerations: The investigators will enroll a total of 120 participants

ELIGIBILITY:
Inclusion Criteria: Breast Cancer Screening Intervention

* Women age 45-75
* Average risk for breast cancer
* Never had a mammogram OR not had a mammogram within the past 2 years
* Residing in the Zuni Pueblo

Exclusion Criteria: Breast Cancer Screening Intervention. Meeting at least one of the following criteria:

* Women with breast implants, pregnant, or breast feeding
* History of breast cancer
* Have new breast complaints such as lump or nipple discharge

Inclusion Criteria: Colorectal Cancer Screening Intervention

* Men and women aged 45-75
* Average risk for colorectal cancer
* Never had a fecal occult blood test (FOBT), or fecal immunochemical test (FIT) or a colonoscopy OR not had a FOBT or FIT in the past year, OR no colonoscopy in the past 10 years
* Residing in the Zuni Pueblo

Exclusion Criteria: Colorectal Cancer Screening Intervention. Meeting at least one of the following criteria:

* History of colorectal cancer, total colectomy, adenomatous polyps, or inflammatory bowel disease
* Up-to-date with colorectal cancer screening
* Severe comorbidity
* Incarceration
* Family history of colorectal cancer
* Hospice/terminal care status

Inclusion Criteria: Cervical Cancer Screening Intervention

* Women aged 21-65
* Never had a cytology (Pap smear) OR had a Pap smear more than 3 years ago OR women aged 30-75, and never had screening with a combination of cytology and human papillomavirus testing OR no combination of testing in the past 5 years
* Residing in the Zuni Pueblo

Exclusion Criteria: Cervical Cancer Screening Intervention. Meeting at least one of the following criteria:

* History of total hysterectomy
* High risk for cervical cancer due to suppressed immune system (e.g., HIV infection, organ transplant, long-term steroid use)
* Women over age 65 who have had regular screenings with normal results

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shiraz I Mishra, MBBS, PhD, Principal Investigator — University of New Mexico School of Medicine
Locations (1):
- University of New Mexico - Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For Aim 3 (Focus Groups, Descriptive): Enrollment n=96, For Aim 4 (Community Survey, Descriptive): Enrollment n=281 For Aim 8 (INT, Pilot Test), recruited 131 participants who had expressed interest to participate in the pilot test of the 3 cancer-specific INTs. The recruitment, followed by the baseline (pre-INT) survey, the 3 cancer-specific INTs, and the post-INT, were conducted between December 2022 and April 2023. Convenience sampling methods were used to recruit the participants
Pre-assignment Details: For Aim 3: Recruitment n=96, For Aim 4: Recruitment n=281, For Aim 8 (INT, Pilot Test), out of the 131 participants enrolled, 117 participants completed all Aim 8 study activities (pre- and post-INT surveys, educational and behavioral INT(s)). Preliminary data on these 117 participants are reported herein. The Zuni Pueblo's Tribal leadership has approved the findings for their wider dissemination. Aims 1, 2, 5, 6, and 7 were descriptive in nature, with no data collection.
Groups:
- Aim 3, Focus Group, Descriptive: Cancer Control Needs: The investigators conducted 12 focus groups to document cancer control needs
- Aim 4, Community Survey, Descriptive: The investigators surveyed adults to document cancer control needs and existing cancer-screening practices
- Aim 8, INT, Pilot Test: Breast, Colorectal, and Cervical Cancer Screening: Breast, Colorectal, and Cervical Cancer Screening Interventions (Aim 8, INT, Pilot Test): The experimental arm comprised of adult men and women divided in three gender/age strata, based on gender/age-specific recommended cancer screening practices. Women age 50-75 years received the interventions for breast, colorectal, and cervical cancers screening. Men age 50-75 years received the intervention for colorectal cancer screening. Women age 21-49 years received the intervention for cervical cancer screening.
Period: Overall Study
Arm/Group | Aim 3, Focus Group, Descriptive: Cancer Control Needs | Aim 4, Community Survey, Descriptive | Aim 8, INT, Pilot Test: Breast, Colorectal, and Cervical Cancer Screening
Started | 96 | 281 | 131
Completed | 96 | 281 | 117
Not Completed | 0 | 0 | 14

BASELINE CHARACTERISTICS:
Groups:
- Aim 3, Focus Groups, Descriptive: Cancer Control Needs: Trained focus group facilitators conducted the focus groups. Each session lasted approximately two hours. The facilitators used a semi-structured focus group guide to explore needs around cancer prevention and control, including knowledge, barriers and support, and communications. Conducted 11 focus groups with Community members (Community, N=85) and 1 focus group with providers (Provider, N=11)
- Aim 4, Community Survey, Descriptive: Cancer Control Needs: The study team conducted surveyed interested participants on their cancer screening practices. The surveys were age/gender specific. Women ages 50-75 were surveyed on breast, cervical, and colorectal cancers. Women aged 21-49 were surveyed on cervical cancer. Men aged 50-75 were surveyed on colorectal cancer
- Aim 8, INT, Pilot Test: Breast, Colorectal, and Cervical Cancer Screening: For Aim 8 (INT Pilot Test), the investigators will train Community Health Representatives (CHRs) in interactive group discussions techniques. CHRs will administer 1 session/week, lasting approximately 2 hours, and conducted among 12 men or women ages 21-75 per cluster. The CHRs will distribute the cancer-specific (i.e., breast, colorectal, and cervical) small media during the first session and refer to it during the course of the 4 sessions. During the sessions, the CHRs will function as a facilitator linking information with practical skills. At the end of the 4-week INT, participants will receive a voucher to present to a designated point-person at the health center who would schedule the screening for the age- and gender-specific cancers.
  Breast, Colorectal, and Cervical Cancer Screening Interventions (Aim 8, INT, Pilot Test): Women age 50-75 years will receive the interventions for breast, colorectal, and cervical cancers screening. Men age 50-75 years will receive the intervention for colorectal cancer screening. Women age 21-49 years will receive the intervention for cervical cancer screening. The 4-week interventions, delivered once a week, will consist of educational sessions that discuss cancer-specific information (i.e., breast, colorectal, and cervical cancer): breast (colorectal, cervical) cancer myths and facts, risk factors and symptoms, screening, and review/action plan. The educational sessions will be complemented by cancer-specific small media (brochure).
- Total: Total of all reporting groups
Arm/Group | Aim 3, Focus Groups, Descriptive: Cancer Control Needs | Aim 4, Community Survey, Descriptive: Cancer Control Needs | Aim 8, INT, Pilot Test: Breast, Colorectal, and Cervical Cancer Screening | Total
Number analyzed (Participants) | 96 | 281 | 117 | 494
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 85 | 226 | 102 | 413
  >=65 years | 11 | 55 | 15 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 171 | 72 | 304
  Male | 35 | 110 | 45 | 190
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 83 | 281 | 117 | 481
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 0 | 0 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Aim 3, Focus Groups, Descriptive: Knowledge, Barriers and Support, and Communication About Breast, Cervix, and Colorectal Cancers
Description: The focus group discussion documents the participants' knowledge about, barriers and support for, and communications about cancer and cancer prevention. Focus group methodology is primarily a qualitative research method and directly quantifying themes is not the typical approach. In this research, only qualitative data were collected with no quantification other than of the number of participants that endorsed a particular theme
Time Frame: 12 months
Population: The number analyzed in each row is based on the total number of participants (Community N=85 in 11 focus groups; Providers N=11 in one focus group) who took part in the focus group sessions
Measure: Count of Participants; unit: Participants
Groups:
- Aim 3, Focus Groups, Descriptive Cancer Control Needs: For Aim 3 (Focus Groups, Descriptive), the investigators will conduct focus groups among Zuni adults and healthcare providers practicing at the Zuni Community Health Center. Through the focus group discussions, the investigators will document cancer control needs in the Zuni Pueblo. The focus group discussion followed a semi-structured format, with stem questions followed up with probes, as needed.
Arm/Group | Aim 3, Focus Groups, Descriptive Cancer Control Needs
Number analyzed (Participants) | 96
Participants
  Knowledge (Community): Variable knowledge and awareness regarding cancer and screening: number analyzed (Participants) | 85
  Knowledge (Community): Variable knowledge and awareness regarding cancer and screening | 85
  Knowledge (Community): Need information about cancers, screening tests, and prevention: number analyzed (Participants) | 85
  Knowledge (Community): Need information about cancers, screening tests, and prevention | 85
  Knowledge (Community): Range of views regarding causality: number analyzed (Participants) | 85
  Knowledge (Community): Range of views regarding causality | 85
  Knowledge (Community): Receptivity to preventive strategies: number analyzed (Participants) | 85
  Knowledge (Community): Receptivity to preventive strategies | 85
  Knowledge (Provider): Low screening due to individual-/system-level barriers: number analyzed (Participants) | 11
  Knowledge (Provider): Low screening due to individual-/system-level barriers | 11
  Barriers/Support (Community): Systemic barriers: number analyzed (Participants) | 85
  Barriers/Support (Community): Systemic barriers | 85
  Barriers/Support (Community): Confidentiality concerns: number analyzed (Participants) | 85
  Barriers/Support (Community): Confidentiality concerns | 85
  Barriers/Support (Community): Benefits of supportive elements to promote better health: number analyzed (Participants) | 85
  Barriers/Support (Community): Benefits of supportive elements to promote better health | 85
  Barriers/Support (Provider): Fear/denial, fatalism, and procrastination: number analyzed (Participants) | 11
  Barriers/Support (Provider): Fear/denial, fatalism, and procrastination | 11
  Barriers/Support (Provider): Social determinants of health: number analyzed (Participants) | 11
  Barriers/Support (Provider): Social determinants of health | 11
  Barriers/Support (Provider): Competing priorities and social conditions: number analyzed (Participants) | 11
  Barriers/Support (Provider): Competing priorities and social conditions | 11
  Barriers/Support (Provider): Systems-level barriers: number analyzed (Participants) | 11
  Barriers/Support (Provider): Systems-level barriers | 11
  Communication (Community): Discuss cancer screening with family: number analyzed (Participants) | 85
  Communication (Community): Discuss cancer screening with family | 85
  Communication (Community): Confidence, trust, gender concordance eases communications: number analyzed (Participants) | 85
  Communication (Community): Confidence, trust, gender concordance eases communications | 85
  Communication (Community): Cultural traditions, gender norms, privacy concern preclude communication: number analyzed (Participants) | 85
  Communication (Community): Cultural traditions, gender norms, privacy concern preclude communication | 85
  Communication (Community): Systems-level factors preclude healthcare discussions: number analyzed (Participants) | 85
  Communication (Community): Systems-level factors preclude healthcare discussions | 85
  Communications (Provider): Prioritize communication about cancer screening: number analyzed (Participants) | 11
  Communications (Provider): Prioritize communication about cancer screening | 11
  Communications (Provider): Aware about screening but not going through it: number analyzed (Participants) | 11
  Communications (Provider): Aware about screening but not going through it | 11
  Communications (Provider): Utilize culturally tailored counseling strategies: number analyzed (Participants) | 11
  Communications (Provider): Utilize culturally tailored counseling strategies | 11
  Communications (Provider): Use humor: number analyzed (Participants) | 11
  Communications (Provider): Use humor | 11
Statistical Analysis 1: Comparison: Aim 3, Focus Groups, Descriptive Cancer Control Needs; All focus groups were summarized together and, therefore, the denominators (N=85 [Community], N=11 [Provider]) for each theme are the same. Further, the focus groups only made qualitative (and no quantitative) assessments/endoresement of themes. No formal comparisons among groups were made; Test type: Other — This is a summary of the total number of participants in the focus groups who endorsed the particular theme; Proportion endorsing themes = 1.0

2. Primary Outcome: Aim 4, Community Survey, Descriptive: Cancer Control Needs
Description: Age/gender specific self-reported screening behaviors for breast, colorectum, and cervical cancers
Time Frame: 7 months
Population: The Number Analyzed in each row reflects the number of participants assessed, while the values reported in the data fields reflect the number of participants who Ever Had the respective screening examinations
Measure: Count of Participants; unit: Participants
Groups:
- Aim 4, Community Survey, Descriptive: Cancer Control Needs: For Aim 4, the investigators will administer eligible participants a survey over the phone. The surveys will document cancer control needs in the Pueblo. The surveys collected data on cancer screening practices
Arm/Group | Aim 4, Community Survey, Descriptive: Cancer Control Needs
Number analyzed (Participants) | 281
Participants
  Ever Had A Mammogram To Screen For Breast Cancer, Women 50-75 years: number analyzed (Participants) | 110
  Ever Had A Mammogram To Screen For Breast Cancer, Women 50-75 years | 95
  Ever Completed an FOBT or Colonoscopy To Screen For Colorectal Cancer, Men and Women 50-75 years: number analyzed (Participants) | 218
  Ever Completed an FOBT or Colonoscopy To Screen For Colorectal Cancer, Men and Women 50-75 years | 92
  Ever Had a Pap Test and/or HPV Test To Screen For Cervical Cancer, Women 21-75 years: number analyzed (Participants) | 171
  Ever Had a Pap Test and/or HPV Test To Screen For Cervical Cancer, Women 21-75 years | 129

3. Primary Outcome: Aim 8, INT, Pilot Test: Age/Gender-specific Breast, Colorectal, and Cervical Cancer Screening
Description: Self-reported receipt of a screening exam, or scheduling an appointment for a screening exam, or self-reported attempt to make an appointment for a screening exam. Cancer-specific screening exams included FOBT/FIT/Colonoscopy for colorectal cancer for men and women 45-75 years, Pap smear for cervical cancer for women 21-75 years, or mammogram for breast cancer for women 45-75 years
Time Frame: 8 months
Population: The number analyzed in each row is based on age/gender strata and the respective cancer screening test. Men and women age 45-75 were eligible for colorectal cancer screening test. Women age 45-75 were eligible for breast cancer screening test, women 21-75 were eligible for cervical cancer screening test.
Measure: Count of Participants; unit: Participants
Groups:
- Breast, Colorectal, and Cervical Cancer Screening (Aim 8, INT, Pilot Test): The study staff will administer to eligible participants the pre-INT and post-INT surveys. The post-INT surveys will be administered approximately 8 months after delivering the INTs. The participants will receive the INT(s) immediately after completing the pre-INT surveys.
  Breast, Colorectal, and Cervical Cancer Screening Interventions (Aim 8, INT, Pilot Test): Adult men and women will receive age- and gender-specific INTs. Women age 45-75 years will receive the interventions for breast, colorectal, and cervical cancers screening. Men age 45-75 years will receive the intervention for colorectal cancer screening. Women age 21-49 years will receive the intervention for cervical cancer screening. The cognitive-behavioral INTs on age-gender specific cancers will range from 1-2 hours. The study team will utilize a digital flipchart that will cover each cancer's specific risk/protective factors, incidence, mortality, screening methods, and resources. The study team member delivering the INTs will function as a facilitator linking information with practical skills.
Arm/Group | Breast, Colorectal, and Cervical Cancer Screening (Aim 8, INT, Pilot Test)
Number analyzed (Participants) | 117
Participants
  Stool Test, Men, 45-75 years (Aim 8, INT, Pilot Test): number analyzed (Participants) | 45
  Stool Test, Men, 45-75 years (Aim 8, INT, Pilot Test) | 20
  Stool Test, Women, 45-75 years (Aim 8, INT, Pilot Test): number analyzed (Participants) | 50
  Stool Test, Women, 45-75 years (Aim 8, INT, Pilot Test) | 28
  Colonoscopy, Men, 45-75 years (Aim 8, INT, Pilot Test): number analyzed (Participants) | 45
  Colonoscopy, Men, 45-75 years (Aim 8, INT, Pilot Test) | 11
  Colonoscopy, Women, 45-75 years (Aim 8, INT, Pilot Test): number analyzed (Participants) | 50
  Colonoscopy, Women, 45-75 years (Aim 8, INT, Pilot Test) | 15
  Mammogram, Women, 45-75 years (Aim 8, INT, Pilot Test): number analyzed (Participants) | 50
  Mammogram, Women, 45-75 years (Aim 8, INT, Pilot Test) | 26
  Pap Smear, Women, 45-75 years (Aim 8, INT, Pilot Test): number analyzed (Participants) | 50
  Pap Smear, Women, 45-75 years (Aim 8, INT, Pilot Test) | 23
  Pap Smear, Women, 21-44 years (Aim 8, INT, Pilot Test): number analyzed (Participants) | 22
  Pap Smear, Women, 21-44 years (Aim 8, INT, Pilot Test) | 21
Statistical Analysis 1: Comparison: Breast, Colorectal, and Cervical Cancer Screening (Aim 8, INT, Pilot Test); Test type: Other — Formal statistical comparisons were not made; Proportion endorsing attempt to screen = 0.567, 95% CI 2-sided [0.303 to 0.831] — Pooled estimate of attempt to screening. Using R: n1 <- c(20,28,11,15,26,23,21); nt <- c(45,50,45,50,50,50,22) p1 <- n1/nt; v1 <- p1*(1-p1)/nt fit <- lm(p1 ~ 1,weight=1/v1) summary(fit)$coef[1] + qt(.975,6)*c(0,-1,1)*summary(fit)$coef[2]

ADVERSE EVENTS:
Time Frame: For Aim 3, t=12 months For Aim 4, t=7 months For Aim 8, t=8 months
Groups:
- Aim 3, Focus Groups, Descriptive: Trained focus group facilitators conducted the focus groups. Each session lasted approximately two hours. The facilitators used a semi-structured focus group guide to explore needs around cancer prevention and control, including knowledge, barriers and support, and communications
- Aim 4, Community Survey, Descriptive: The study team conducted surveyed interested participants on their cancer screening practices. The surveys were age/gender specific. Women ages 50-75 were surveyed on breast, cervical, and colorectal cancers. Women aged 21-49 were surveyed on cervical cancer. Men aged 50-75 were surveyed on colorectal cancer
- Aim 8, INT, Pilot Test: The study staff will administer to eligible participants the pre-INT and post-INT surveys. The post-INT surveys will be administered approximately 8 months after delivering the INTs. The participants will receive the INT(s) immediately after completing the pre-INT surveys.
  Breast, Colorectal, and Cervical Cancer Screening Interventions: Adult men and women will receive age- and gender-specific INTs. Women age 45-75 years will receive the interventions for breast, colorectal, and cervical cancers screening. Men age 45-75 years will receive the intervention for colorectal cancer screening. Women age 21-49 years will receive the intervention for cervical cancer screening. The cognitive-behavioral INTs on age-gender specific cancers will range from 1-2 hours. The study team will utilize a digital flipchart that will cover each cancer's specific risk/protective factors, incidence, mortality, screening methods, and resources. The study team member delivering the INTs will function as a facilitator linking information with practical skills.
Arm/Group | Aim 3, Focus Groups, Descriptive | Aim 4, Community Survey, Descriptive | Aim 8, INT, Pilot Test
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/281 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/281 | 0/117
Other Adverse Events (participants affected / at risk) | 0/96 | 0/281 | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT04259762/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT04259762/ICF_001.pdf